CLINICAL TRIAL: NCT03743337
Title: Study of Coaching Practices in Early Care and Education Settings
Acronym: SCOPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Child Trends (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Other Study IDs: 50320
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Early Childhood Professional Development
Keywords: Infant-toddler care; Early child development; Professional development

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mathematica Policy Research, funded by the Administration for Children and Families (ACF) in the U.S. Department of Health and Human Services (HHS) will collect descriptive information for the Study of Coaching Practices in Early Care and Education Settings (SCOPE) project. The goal of this information collection is to learn how the prevalence, implementation, combination, and tailoring of core features of professional development coaching for early care and education (ECE) providers vary across ECE classrooms and family child care (FCC) homes serving children supported by Child Care and Development Fund (CCDF) subsidies or in settings that receive Head Start grants. The investigators will conduct three data collection activities. First, the investigators will collect information on coaching taking place in different states in winter 2018 from state-level entities. Second, the investigators will conduct one round of survey data collection with ECE center directors, coaches, teachers, and FCC providers in winter 2019 through spring 2019. Third, the investigators will conduct case studies to better understand factors that influence the coaching approaches identified through the survey data collection. The case studies will include semi-structured interviews, a coaching session observation, and collection of coaching logs. The case studies will occur in spring 2020.

DETAILED DESCRIPTION:
This study aims to advance understanding of implementation of core features of coaching in ECE classrooms, and how features may vary by key contextual factors and implementation drivers. This study will focus on coaching used for delivering professional development services to ECE teachers and FCC providers to improve knowledge and practice in center-based classrooms and FCC homes serving preschool-age children. At the classroom/teacher level, the approach to coaching can vary by dosage, content, activities (e.g., assessment, observation, goal-setting, modeling, reflection), materials (e.g., video, written plans, resource documents) and other features. However, there is no consensus as to which of these features are core to the practice of coaching. Additionally, little is known about how these features of coaching are implemented, combined, and tailored to the needs of teachers or how contextual factors or implementation drivers may mediate or moderate the effects of coaching. Ultimately, SCOPE findings will improve coaching practice in the ECE field and determine which coaching features are ripe for more rigorous evaluation.

Descriptive Study: The investigators will carry out a descriptive study in a sample of seven states. Sampled states will have one or more classroom-based coaching models offered to centers and FCC homes that are serving preschool-age children and that receive Head Start grants or serve children who receive CCDF subsidies. All of the data that will be collected are listed below.

1. State coaching informant interviews: To obtain information about coaching approaches and about the available administrative data on coaching, including the range of coaching providers and approaches occurring in states and what ECE settings may be receiving classroom coaching. As part of this process, we will also seek existing administrative data on coaching processes and participants.
2. ECE setting eligibility screening: To obtain information on the characteristics of the ECE setting, the coaching taking place in that setting, and characteristics of participants in coaching; and to determine if a setting is eligible for survey data collection and if personnel are willing to participate in the study
3. Surveys for the descriptive study:

   * A center director survey - To collect information on the center context, supports for and challenges to coaching and professional development, and structural and process features of coaching
   * A coach survey - To collect information on coach characteristics, supports for and challenges to coaching, and process and structural features of coaching
   * A teacher/FCC provider survey- To collect information on teacher and FCC provider characteristics, supports for coaching, structural and process features of coaching, coaching outputs (such as attitudes and beliefs), and the FCC context

Case Studies: The investigators will also conduct case studies in twelve ECE settings (centers and FCC homes) selected from the seven states; some of the settings may have participated in the descriptive study and others may not have. Site visit data collection for the case studies will consist of the following activities:

1. Semi-structured interviews with center directors, teachers/FCC providers, coaches, and coach supervisors. To collect information on how decisions are made about coaching and what features are included; supports for coaching; organizational context and climate for coaching (e.g., organizational culture, philosophies, staffing and turnover, languages and cultures of families served); individual experiences as part of the coaching process; barriers/supports for coaching
2. Teacher/FCC provider survey: The teachers and FCC providers in the case studies will be asked to complete the descriptive study teacher/FCC provider survey.
3. Collection of coaching logs (whenever available): To provide information on the frequency of interactions between teachers/FCC providers and coaches, the focus of these interactions, and the coaching strategies employed. The coaching logs are preexisting materials used by some coaches when they provide coaching to teachers.
4. Coaching session observations: To provide information on the process features of coaching (coaching activities and relationship-building activities); structural features (target of coaching and content); and outputs (teacher/FCC provider engagement, actual dosage, and perceptions of the coach-teacher/FCC provider relationship)

ELIGIBILITY:
Inclusion Criteria:

1. Currently operating licensed or license exempt child care setting
2. Receiving funding from a Head Start grant and/or serve children who receive CCDF subsidies
3. Currently receiving classroom-based coaching for teachers of preschoolers/FCC providers caring for preschoolers.

Exclusion Criteria:

* Does not meet the inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Early care and education (ECE) center directors, professional development coaches and coach supervisors, center-based teachers, and family child care (FCC) providers.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-06-21 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Coaching experienced by teachers/family child care providers | Up to 6 months
  Study-developed teacher/FCC provider survey on coaching experiences
Coaching delivered by professional development coaches | Up to 6 months
  Study developed survey of coaches' approach to coaching
Context in which coaching takes place/influences on the coaching process | Up to 6 months
  Study developed survey of center directors on center characteristics
Director perspectives external factors that influence the implementation of coaching | Up to 3 months
  Study developed interview of center directors on program and system level contextual factors that influence coaching
Coaching participant perspectives on external factors that influence the implementation of coaching | Up to 3 months
  Study developed interview of teachers/FCC providers
Coach perspectives on external factors that influence the implementation of coaching | Up to 3 months
  Study developed interview of coaches on program and system level contextual factors that influence coaching
Coach supervisor perspectives on external factors that influence the implementation of coaching | Up to 3 months
  Study developed interview of coach supervisors on program and system level contextual factors that influence coaching
Content of coaching interactions | Up to 90 minutes
  Study developed observation of coach-teacher/FCC provider professional development coaching sessions

CONTACTS AND LOCATIONS:
Overall Officials: Emily Moiduddin, PhD, Study Director — Mathematica Policy Research; Sally Atkins-Burnett, PhD, Principal Investigator — Mathematica Policy Research
Locations (1):
- Mathematica, Washington D.C., District of Columbia, United States